CLINICAL TRIAL: NCT06857110
Title: "Supracondylar Radial Nerve Block Guided by Ultrasound Versus Hematoma Block for Analgesic Management in Closed Reduction of Distal Radius Fractures: a Randomized Controlled Clinical Trial"
Brief Title: "Supracondylar Radial Nerve Block Guided by Ultrasound Versus Hematoma Block for Analgesic Management in Closed Reduction of Distal Radius Fractures"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario San Ignacio (Other)
Collaborators: Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Distal Radius Fracture
Keywords: Wrist fractures; closed fracture reduction; analgesia; Anesthesia, local; nerve block; pain measurement
MeSH Terms: conditions — Wrist Fractures; Agnosia

STUDY DESIGN:
Masking Description: No masking Since this study involves two non-invasive, clearly distinguishable interventions, it is not possible to blind the patient to the assigned treatment or to blind the healthcare professionals administering the intervention or recording the outcome. However, data analysis will be conducted with blinding of the administered intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hematoma block (Active Comparator): The orthopedic surgeon on duty will perform the hematoma block prior to closed reduction in the procedure room as follows: 75 mg of intramuscular diclofenac will be administered, or 1 gram of oral acetaminophen in case of contraindications for the administration of Non-Steroidal Anti-inflammatory Drugs.
  With the patient in supine position, palpation will be conducted to locate the fracture. The skin above this area will be cleaned with 2% chlorhexidine gluconate antiseptic solution and sterile gauze. While wearing sterile gloves, the orthopedic surgeon will insert a 10 cc syringe with a 21 gauge needle and aspirate to confirm placement over the fracture hematoma. 1% Lidocaine without epinephrine will be infiltrated (dose of 2mg/kg). A 10-minute waiting period will be observed before performing closed reduction maneuvers.
  Interventions: Procedure: hematoma block; Drug: 5 mg of intramuscular diclofenac
- Procedure/surgery (Experimental): The orthopedic surgeon will perform an ultrasound-guided supracondylar block of the radial nerve prior to closed reduction. Intramuscular diclofenac (75 mg) or oral acetaminophen (1 g) will be administered if NSAIDs are contraindicated. With the patient seated, the lateral epicondyle of the humerus will be identified through palpation and ultrasound. After antisepsis with 2% chlorhexidine gluconate, a non-cutting needle (Stimuplex 50 mm) will be inserted approximately 3 cm proximal to the lateral epicondyle, and 1% lidocaine (2 mg/kg) without epinephrine will be administered. A 10-minute waiting period will be observed before performing the closed reduction maneuvers.
  Interventions: Procedure: ultrasound-guided supracondylar block of the radial nerve

INTERVENTIONS:
Procedure: ultrasound-guided supracondylar block of the radial nerve — 75 mg of intramuscular diclofenac will be administered, or 1 gram of oral acetaminophen in case of contraindications for the administration of Non-Steroidal Anti-inflammatory Drugs
  Arms: Procedure/surgery
Procedure: hematoma block — The orthopedic surgeon will perform a hematoma block before closed reduction. Intramuscular diclofenac (75 mg) or oral acetaminophen (1 g) will be administered if NSAIDs are contraindicated. With the patient in a supine position, the fracture site will be identified through palpation. After antisepsis with 2% chlorhexidine gluconate, a 10 cc syringe with a 21-gauge needle will be inserted to aspirate and confirm placement over the fracture hematoma. Then, 1% lidocaine (2 mg/kg) without epinephrine will be infiltrated. A 10-minute waiting period will be observed before performing closed reduction maneuvers.
  Arms: hematoma block
Drug: 5 mg of intramuscular diclofenac — the orthopedic surgeon on duty will perform the hematoma block prior to closed reduction in the procedure room as follows: 75 mg of intramuscular diclofenac will be administered
  Arms: hematoma block

SUMMARY:
Non-surgical treatment with closed reduction and immobilization using a splint or cast is the preferred approach for stable distal radius fractures, particularly in elderly patients. It is also the initial intervention for displaced fractures with a surgical indication before the procedure, aiming to reduce edema, manage pain, and prevent associated complications. However, the maneuvers required for bone reduction can cause significant pain, and there is still insufficient evidence to favor one anesthetic method over another. In recent years, there has been a trend toward utilizing local methods, such as hematoma block or ultrasound-guided supracondylar block of the radial nerve, due to their lower incidence of complications. Nonetheless, there are currently no studies comparing the efficacy of these two analgesic approaches.

This study aims to compare the analgesic effect of ultrasound-guided supracondylar block with that obtained through hematoma block in patients with distal radius fracture during closed reduction, using the Numeric Rating Scale. Additionally, it aims to compare the quality of the reduction through radiographic measures and assess the frequency of adverse events after the two interventions.

DETAILED DESCRIPTION:
Approval has been obtained from the ethics committee. A process of informed consent will be conducted with all participants, ensuring confidentiality and data protection. Once the informed consent is signed, either an orthopedic surgeon or resident will gather demographic data such as age, sex, height, weight and analgesics taken during the same day of the intervention. Additionally, the type of fracture according to the AO classification and the perceived pain before the intervention will be registered in REDCap

Subsequently, this healthcare personnel in the emergency room will contact a member of the research team, who will conduct randomization of the intervention though REDcap and determine which analgesic approach should be offered to the participant.

Training and education will be provided to orthopedic surgeons working in the emergency room to standardize the local analgesic interventions, following the recommendations outlined in the study protocol.

Since this study involves two non-invasive, clearly distinguishable interventions, it is not possible to blind the patient to the assigned treatment or to blind the healthcare professionals administering the intervention or recording the outcome. However, data analysis will be conducted with blinding of the administered intervention.

After a 10-minute waiting period following the analgesic procedure, the participants' pain will be reassessed using the numeric pain scale. After this, all patients will undergo closed reduction through manual reduction maneuvers. This involves the patient being placed in supine position, while two doctors perform traction along the axis of the arm and countertraction at the elbow for 2-5 minutes to impact the fracture. Subsequently, wrist extension, flexion, and ulnar deviation of at least 15° will be performed, with manual pressure applied on the dorsal aspect of the radius if necessary. Finally, the patient will be immobilized with a brachy metacarpal closed cast or splint, and post-reduction radiographs will be taken. Patients will be asked to rate the pain experienced during this reduction.

Radiographs before and after the reduction will also be taken, following a standardized protocol. The posteroanterior projection will be performed with the wrist and elbow at shoulder height, aligning the joints in the transverse plane. The palm of the hand will be in contact with the cassette, as in this position, the radius and ulna are parallel. The lateral projection will be taken with the shoulder, elbow, and wrist aligned in the sagittal plane, positioning the edge of the distal ulna on the cassette. In the posteroanterior projection, the radial height, ulnar variance, and radial inclination will be measured, while the dorsal/volar tilt will be measured on the lateral projection.

Finally, all complications during the procedure or adverse effects occurring 3 hours after the intervention will be registered.

An intention-to-treat analysis will be conducted. Descriptive statistics will be generated using R studio for the demographic variables. The proportion of patients experiencing a reduction greater than two points (which corresponds to the minimal clinically important difference) between baseline pain and pain experienced after the analgesic procedure and during the reduction will be registered and compared using an exact Fischer test.

Additionally, the proportion of patients with an adequate reduction will be compared between the two interventions for each of the radiographic measures, categorized as within or outside the ideal range. Finally, the proportion of complications and adverse effects for each intervention will be compared using an exact Fischer test.

An interim analysis will be conducted when half of the sample has been recruited to evaluate the efficacy and safety of the interventions in a blinded manner. The study will conclude if clear benefits are found with an intervention or if statistically significant harm is evidenced. An O'Brien-Fleming method will be employed to adjust the significance level for this interim analysis, aiming to control Type I error.

The results will be reported collectively for publication in a peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old with skeletal maturity evidenced in the initial radiographs.
* Patients with a radiological diagnosis of distal radius fracture
* Patients whose clinical condition is considered acute (duration of symptoms less than one week).
* Patients who have an indication for closed reduction as a definitive or initial management of their distal radius fracture
* Patients treated at San Ignacio University Hospital in Bogotá, Colombia

Exclusion Criteria:

* • Patients with bilateral distal radius fractures

  * Patients with open distal radius fractures.
  * Patients with another fracture in the same limb
  * Patients in a state of intoxication or under the influence of psychoactive substances.
  * Patients with hemodynamic instability that prevents prioritizing closed reduction as management.
  * Patients with a known allergy to local anesthetics
  * Patients on full-dose anticoagulant therapy.
  * Patients who refuse to participate in the study
  * Patients with cognitive, visual, or auditory impairments that prevent the proper completion of questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain during closed | Approximately 30 minutes after the patient's arrival at the orthopedic emergency department and 15 minutes after the analgesic intervention
  Pain experienced during the closed reduction of the distal radius fracture, measured by the numeric pain scale and reported immediately after the reduction maneuvers

SECONDARY OUTCOMES:
Pain reduction after the analgesic procedure | Approximately 15 minutes after the patient's arrival at the orthopedic emergency department
  Proportion of patients experiencing a reduction greater than two points (which corresponds to the minimal clinically important difference) between baseline pain and pain experienced after the analgesic procedure. the escale use is Visual Analogue Scale. It consists of a horizontal line of 10 cm (or 100 mm), where one end represents "no pain" (0) and the other end "the worst pain imaginable" (10 or 100, depending on the scale used). The higher the scale value, the worse the patient's health condition and the greater the pain.
Pain reduction measured after the closed reduction | : Approximately 30 minutes after the patient's arrival at the orthopedic emergency department and 15 minutes after the analgesic intervention
  proportion of patients experiencing a reduction greater than two points (which corresponds to the minimal clinically important difference) between baseline pain and during the closed reduction of the fracture
quality of reduction measured by dorsal tilt | Approximately 45 minutes after the patient's arrival at the orthopedic emergency department
  in a lateral x-ray wrist projection, dorsal tilt is the angle formed between a line drawn between the most distal points of the dorsal and palmar lips of the distal radius and a line perpendicular to the axis of the radius. This measurement is important as its value is directly associated with the functional position of the wrist and its extension capacity. Its alteration is related to a dorsal displacement of the contact surface between the radius, scaphoid, and lunate, causing an abnormal increase in joint pressure and dysfunction of radiocarpal stability. It has been established that a volar tilt of less than 3° after reduction is inadequate.
quality of reduction measured by radial inclination | Approximately 45 minutes after the patient's arrival at the orthopedic emergency department
  In a posteroanterior x-ray wrist projection, radial inclination is the angle between a line drawn from the styloid tip to the lunate facet of the radius and a line perpendicular to the axial axis of the radius. Its normal value i son average 21 to 25 degrees.
quality of reduction measured by radial height | Approximately 45 minutes after the patient's arrival at the orthopedic emergency department
  In a posteroanterior x-ray wrist projection,radial height is the distance between a tangent from the tip of the radial styloid process and a tangent from the most distal part of the ulnar head. This measurement is important as it has been shown that shortening of the distal radius leads to an increase in load at the ulna level, resulting in post-traumatic arthritis, as well as alteration of load transmission leading to degenerative changes in the articular cartilage and changes in wrist stability. It has been described that a radial height less than 9.3 mm is inadequate if present after reduction
quality of reduction measured by ulnar variance | Approximately 45 minutes after the patient's arrival at the orthopedic emergency department
  : In a posteroanterior x-ray wrist projection,ulnar variance is the distance between a line perpendicular to the axis of the radius traced through the distal ulnar aspect of the radius and a line drawn by the distal cortex of the ulna. Its normal value should be between -1 to 1mm.
Complications | Approximately 30 minutes after the patient's arrival at the orthopedic emergency department
  proportion of complications during the execution of the intervention
Adverse events | during the first three hours after the intervention
  Proportion of adverse events during the first three hours after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Luis A García González, Orthopedic Surgeon and Traumat, Principal Investigator — Hospital Universitario San Ignacio
Locations (1):
- Hospital Universitario San Ignacio, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: No